CLINICAL TRIAL: NCT07207512
Title: Emotion-Focused Therapy in the Treatment of Prolonged Grief Disorder: Study Protocol for a Randomised Controlled Trial
Brief Title: Emotion-Focused Therapy in the Treatment of Prolonged Grief Disorder
Acronym: EFT-PGD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia Comillas (Other)
Responsible Party: Principal Investigator, José Gamoneda Larripa, Associate professor, Universidad Pontificia Comillas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPComillas-EFT-PGD
Record Dates: First submitted 2025-09-26; First posted 2025-10-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Prolonged Grief Disorder (PGD)
Keywords: grief; bereavement; prolonged grief disorder; grief with complications; Emotion-Focused Therapy; PGD; Randomized Controlled Trial; RCT; study protocol; Treatment Effectiveness
MeSH Terms: conditions — Prolonged Grief Disorder | interventions — Emotion-Focused Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion-Focused Therapy for Grief (Experimental)
  Interventions: Behavioral: Emotion-Focused Therapy for Grief
- self-help intervention based on Emotion-Focused Therapy (Placebo Comparator)
  Interventions: Behavioral: Self-help intervention based on EFT

INTERVENTIONS:
Behavioral: Emotion-Focused Therapy for Grief — The EFT intervention will follow the model described in EFT for grief. Its main goal is to transform core emotional pain (e.g., chronic shame) by activating change-inducing emotions (e.g., assertive anger), a process described as "changing emotion with emotion." This work takes place within a safe and supportive therapeutic relationship, characterized by the therapist's empathic, accepting, and compassionate stance. Therapists remain attuned to emotional markers (e.g., self-criticism, unfinished business) that signal opportunities for targeted work on specific affective problems, which are usually addressed through experiential tasks such as the Empty-Chair for Unfinished Business. Although EFT is transdiagnostic, grief work has certain distinctive features, such as the central role of experiencing grief-related sadness and fostering a sense of connection with the deceased.
  Arms: Emotion-Focused Therapy for Grief
Behavioral: Self-help intervention based on EFT — The self-help intervention consists of 10 written exercises designed to address different aspects of grief. These include psychoeducation, emotional regulation, focusing on bodily awareness, softening self-criticism, reducing avoidance, managing anxiety and fear, clarifying confusing emotional reactions, processing trauma, imaginal dialogues with the deceased, and cultivating compassion.
  Arms: self-help intervention based on Emotion-Focused Therapy

SUMMARY:
The goal of this clinical trial is to learn if Emotion-Focused Therapy (EFT) works to reduce symptoms of Prolonged Grief Disorder (PGD) in adults. PGD happens when the pain of losing a loved one lasts a long time and causes serious problems in daily life.

* The main questions this study aims to answer are:

  1. Does EFT lower grief symptoms in adults with PGD?
  2. Does EFT also help with related problems, such as anxiety, depression, trauma, and overall distress?
* Who can take part:

Adults (18 years or older) who lost a loved one at least 6 months ago and meet the criteria for PGD.

- What will happen in the study:

Participants will be randomly assigned to one of two groups:

1. EFT group: 8 to 10 weekly, face-to-face therapy sessions with a trained therapist.
2. Self-help group: 10 weekly self-help exercises based on EFT, completed on their own.

   * All participants will complete questionnaires on grief, mood, and well-being before starting, during the study, at the end of treatment (12 weeks), and again at 5 months and 12 months after starting.
   * In the EFT group, the therapeutic relationship will also be measured during sessions 3 and 8.
   * Why this study is important:

Most current treatments for grief are based on cognitive-behavioral therapy, but not everyone benefits from them. EFT is a promising therapy that focuses on emotions and has shown positive results for other mental health problems. This trial will test if EFT can be an effective treatment for people struggling with prolonged grief.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Undergoing a grief process (including perinatal grief).
* Meeting diagnostic criteria for Prolonged Grief Disorder (bereavement occurring six months or more prior to the loss; PG-13-R score ≥30).
* Provision of informed consent.
* Stable psychopharmacological medication for at least six weeks prior to therapy onset, with physician approval to maintain stability during the intervention.

Exclusion Criteria:

* Concurrent psychological treatment
* Bereavement occurring less than six months prior to the loss
* Substance abuse
* Eating disorder
* Psychosis;
* Organic brain syndrome
* Suicide risk
* Risk of harm to others.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Prolonged Grief Scale 13 - Revised | From enrollment to the end of the research at 1 year follow-up
  Higher scores indicate greater symptomatology of Prolonged Grief Disorder; a score of 30 or higher meets the clinical threshold for Prolonged Grief Disorder.

SECONDARY OUTCOMES:
Centrality of Event Scale | From enrollment to the end of the reserch at 1 year follow-up
  Higher scores indicate greater trauma symptomatology
Clinical Outcomes in Routine Evaluation-10 | From enrollment to the end of the reserch at 1 year follow-up
  Higher scores indicate greater psychological distress
Patients Health Questionnarie 9 | From enrollment to the end of the reserch at 1 year follow-up
  Higher scores indicate greater psychological distress
Generalized Anxiety Disorder-7 Scale | From enrollment to the end of the reserch at 1 year follow-up
  Higher scores indicate greater GAD symptomatology

CONTACTS AND LOCATIONS:
Overall Officials: José Gamoneda, PhD, Principal Investigator — Universidad Pontificia Comillas
Locations (1):
- Unidad Clínica de Psicología de la Universidad Pontificia Comillas (UNINPSI), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes